CLINICAL TRIAL: NCT05313633
Title: Efficacy of Plyometric Exercises Versus Wii Training on Upper Extremity Function in Children with Unilateral Cerebral Palsy: a Randomized Controlled Trial
Brief Title: Plyometric Exercises Versus Wii Training in Children with Unilateral Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: plyometric training
Record Dates: First submitted 2022-03-07; First posted 2022-04-06 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2022-12

CONDITIONS: Sports Physical Therapy
Keywords: Cerebral palsy; Unilateral Cerebral Palsy; hand grip strength; upper extremity function; range of motion; Wii training; plyometric exercises
MeSH Terms: conditions — Cerebral Palsy | interventions — Occupational Therapy; Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wii group (Experimental): Children in this group will receive a designed physical therapy and occupational therapy programs
  Interventions: Other: Occupational therapy; Other: Wii training
- plyometric group (Experimental): Children in this group will receive a designed physical therapy and occupational therapy programs and plyometric training
  Interventions: Other: Occupational therapy; Other: Plyometric training

INTERVENTIONS:
Other: Occupational therapy — Both groups received a designed occupational therapy program for 30 minutes
Other: Plyometric training — The designed plyometric training program basically focuses on upper extremity strength training and is developed according to the guidelines of the National Strength and Conditioning Association.
  Arms: plyometric group
Other: Wii training — The dose of Wii training was 40 minutes, three times a week for 12 weeks which is an interactive motion-based device.
  Arms: Wii group

SUMMARY:
Plyometric training includes muscle contraction that moves rapidly from the eccentric to the concentric phase of movement while using proper biomechanics. It is an effective neuromuscular stimulus that can improve motor functions of children with cerebral palsy. In plyometric training, muscles exert maximum force in short intervals of time, with the goal of increasing power.

Commercially available video games have been used for a wide range of clinical populations with generally positive clinical outcomes. They have been shown to be active enough to provide an increase in energy expenditure and physical activity in children with cerebral palsy. Furthermore, an early case study showed improvements in visual-perceptual processing, balance, and mobility in a child with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* aged 8-12 years;
* able to understand and follow simple commands.

Exclusion Criteria:

- severe uncontrolled seizures;

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Upper extremity function | after 3 months of treatment
  The quality of upper extremity skill test is a reliable and valid tool used to measure the motor function in children with cerebral palsy. The total scores for each domain percentage score range from zero to 100%
Hand grip strength | after 3 months of treatment
  The hand held dynamometer (Patterson Medical, Warrenville, IL, USA) is a valid and reliable tool to assess grip strength. Each child performs three trials and the mean will be recorded in kilogram for statistical analysis.

SECONDARY OUTCOMES:
Range of motion | after 3 months of treatment
  An electronic goniometer will be used for the measurements of ROM of the affected upper limb in order to accurately track progress in a rehabilitation program.
  Shoulder flexion and abduction, elbow extension, forearm supination and wrist extension will be measured for all children before and after treatment
Selective motor control | after 3 months of treatment
  Test of arm selective control, a valid and reliable tool, will be used to measure selectivity of upper extremity with total score for each upper extremity is 16 and 32 for both tested upper extremities.

CONTACTS AND LOCATIONS:
Overall Officials: walaa A El-nabie, Phd, Study Chair — Cairo university, faculty of physical therapy; Hazem A Ali, Phd, Study Director — Cairo university, faculty of physical therapy
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No